CLINICAL TRIAL: NCT01605045
Title: Efficacy of Fluoroscopy-save Function During Cardiac Catheterization
Brief Title: Screening for Coronary Artery Disease Using Fluoroscopy During Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, James Slater, Director of Cardiac Catheterization Laboratory, NYU Langone Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S12-00007
Record Dates: First submitted 2012-05-10; First posted 2012-05-24 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac catheterization; Radiation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoroscopy-save group (Experimental): Coronary anatomy visualized under fluoroscopy, documented using the fluoroscopy-save function, and further visualized using cinematography only when higher quality is necessary (fluoroscopy-save technique)versus
  Interventions: Other: Fluoroscopy-save group
- Standard technique (Active Comparator): Coronary anatomy visualized and documented using cinematography alone (standard technique)
  Interventions: Other: Standard technique

INTERVENTIONS:
Other: Fluoroscopy-save group — Coronary anatomy visualized under fluoroscopy, documented using the fluoroscopy-save function, and further visualized using cinematography only when higher quality is necessary (fluoroscopy-save technique) versus Coronary anatomy visualized and documented using cinematography alone (standard technique)
  Arms: Fluoroscopy-save group
Other: Standard technique — Coronary anatomy visualized under fluoroscopy, documented using the fluoroscopy-save function, and further visualized using cinematography only when higher quality is necessary (fluoroscopy-save technique) versus Coronary anatomy visualized and documented using cinematography alone (standard technique)
  Arms: Standard technique

SUMMARY:
The aim of this study is to evaluate the effects of screening using the fluoroscopy-save function on reduction of radiation exposure and quality of angiogram during cardiac catheterization when compared to traditional cinematography-guided coronary angiography.

DETAILED DESCRIPTION:
The study will be a prospective, randomized study of patients undergoing clinically-indicated coronary angiograpy in the New York University (NYU) Langone Medical Center cardiac catheterization laboratory. Patients will be randomized to one of two coronary angiography protocols: (1) Coronary anatomy visualized under fluoroscopy, documented using the fluoroscopy-save function, and further visualized using cinematography only when higher quality is necessary (fluoroscopy-save technique) versus (2) Coronary anatomy visualized and documented using cinematography alone (standard technique). The primary outcome will be a measure of radiation exposure to the patient, surface peak skin dose, as measured by the Gafchromic XR RV3 film strip, which is placed under the patient's back during the procedure. Other outcome measures will include radiation output recorded by the fluoroscopy machine, amount of contrast used, and quality of angiograms performed. To determine if the quality of the angiograms performed using the fluoroscopy-save technique is non-inferior to the standard technique, one extra picture will be taken at random using the mode that the study was not randomized to. For example, in the fluoroscopy-save group, a picture that was not visualized under cinematography during the study will be repeated and documented under cinematograpy. In the standard group, a picture will be repeated and documented using the fluoroscopy-save function. These 2 pictures from each study will then be collated and put together in no particular order with all identifiers removed. These single pictures will be read by 2 interventional cardiologists not involved in the study in a blinded fashion. The degree of coronary artery disease as determined by these 2 readers will be compared between the fluoroscopy-save picture and cinematography picture.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the cardiac catheterization laboratory at the NYU Langone Medical Center.
* Patients will be eligible if they are more than 18 years of age and are referred for coronary angiography.

Exclusion Criteria:

* Patients will be excluded if they have reduced renal function since they must receive as minimal of contrast amount as possible, and if their abdominal circumference is > 45 inches since the quality of images under fluoroscopy alone is poorer in patients with increased abdominal girth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measure of radiation exposure to the patient | During coronary angiography
  Surface peak skin dose, as measured by the Gafchromic XR RV3 film strip, which is placed under the patient's back during the procedure.

SECONDARY OUTCOMES:
Dose area product from coronary angiography system | During coronary angiography
Quality of angiograms
  One extra picture will be taken at random using the mode that the study was not randomized to. These 2 pictures from each study will then be collated and put together in no particular order with all identifiers removed. These single pictures will be read by 2 interventional cardiologists not involved in the study in a blinded fashion and degree of correlation between the fluoroscopy-save picture and cinematography picture will be recorded.
30-day events | 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: James Slater, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States